CLINICAL TRIAL: NCT03945799
Title: A Single Group, Open Label, Multi-center Clinical Study to Assess the Efficacy and Safety of Anlotinib in HCC Patients at High Risk of Post Surgery Recurrence.
Brief Title: A Multicenter Study of Anlotinib in Hepatocellular Carcinoma (HCC) Patients at High Risk of Post Surgery Recurrence
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study has gotten preliminary results and stopped advanced.
Sponsor: Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other); West China Hospital (Other); Huashan Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Hospital of Jilin University (Other); Tianjin First Central Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiao Xu, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KY2019-AHR-ZJU
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Administration Anlotinib and it should be continued until relapse of HCC or intolerable toxicity or patients withdrawal of consent.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib: 12mg QD PO d1-14, 21 days per cycle, 8 cycles.

SUMMARY:
To assess the primary effects and safety of Anlotinib in HCC patients at high risk of post surgery recurrence.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most common malignant tumors in the world with high incidence and mortality. Recurrence of HCC is still a great challenge and threat to the patients after resection surgery. Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR), and c-kit. HCC patients who meet the eligibility criteria of this clinical trial will be administrated Anlotinib 12mg QD PO d1-14, 21 days per cycle. The disease free survival (DFS), overall survival (OS) and any adverse effect during the 8 cycles of Anlotinib treatment will be evaluated in order to assess the primary effects and safety of Anlotinib in HCC patients at high risk of post surgery recurrence.

ELIGIBILITY:
Inclusion Criteria:

* No allergic history of Anlotinib
* 18-75 years
* No history of severe arrhythmia or heart failure
* No history of severe ventilation dysfunction or severe pulmonary infection
* No acute or chronic renal failure, creatinine clearance > 40 mL/min
* Liver function is normal: child-pugh grade A or grade B (≤7 points), total bilirubin ≤ 3.0 mg/dL, albumin ≥ 28 g/L, AST, ALT, ALP≤ 5 times of the upper limit of normal value
* Blood test: the absolute neutrophil count ≥ 1.5×10^9 /L, Hb ≥ 8.5 g/L, PLT ≥ 75×10^9 /L (without blood transfusions and drug therapy 14 days before the screening)
* Blood coagulation function: INR≤2.3
* ECOG: 0-2
* Pathology: hepatocellular carcinoma
* Satisfy any of the following:

A. portal vein, hepatic vein or bile duct carcinoma thrombus B. microvascular invasion (MVI) grade II (> 5 MVI, or MVI occurs in the area more than 1 cm from the tumor) C. tumor number ≥ 3 D. preoperative rupture of tumor or tumor invasion adjacent organs

* Patients participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients who have had or are currently complicated with other malignant tumors
* Recurrent hepatocellular carcinoma
* Patients who participated in other clinical trials within 1 month
* Patients with mental illness
* Patients treated with targeted drugs, immunotherapy (such as PD1 antibody), FOLFOX systemic chemotherapy or huaier granules after surgery
* Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Disease free survival | From randomization to recurrence of HCC or death (up to 1year)
  The period from resection surgery to recurrence of HCC

SECONDARY OUTCOMES:
Adverse effect | Up to 1year
  Any adverse effects occur during the use of anlotinib
Overall survival | 1 year
  The survival rate in a year

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes